CLINICAL TRIAL: NCT02339220
Title: Harnessing Neuroplasticity to Promote Rehabilitation: Constraint-Induced (CI) Therapy for Traumatic Brain Injury (TBI)
Brief Title: The Brave Initiative: Bringing Rehabilitation to American Veterans in an Enriched Environment
Acronym: TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gitendra Uswatte, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PT130232
Record Dates: First submitted 2015-01-08; First posted 2015-01-15 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Traumatic Brain Injury
Keywords: Constraint-Induced Movement Therapy; Physical Therapy; Rehabilitation; Occupational Therapy; Fitness Training; Recovery of Function; Neuroplasticity; Exercise Therapy; Brain Injuries; Traumatic Brain Injury; Physical Therapy Modalities; Neuroimaging
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard CI Therapy Group (Experimental): This group will receive Constraint-Induced Movement Therapy (CIMT) with the Standard Transfer Package (sTP).
  Interventions: Behavioral: Constraint-Induced Movement Therapy (CIMT); Behavioral: standard Transfer Package (sTP)
- Enhanced CI Therapy Group (Experimental): This group will receive CIMT with the enhanced Transfer Package (eTP).
  Interventions: Behavioral: Constraint-Induced Movement Therapy (CIMT); Behavioral: enhanced Transfer Package (eTP)
- Standard Fitness Training Group (Active Comparator): This group will receive Lakeshore Enriched Fitness Training (LEFT) with the standard Transfer Package (sTP).
  Interventions: Behavioral: Lakeshore Enriched Fitness Training (LEFT); Behavioral: standard Transfer Package (sTP)
- Enhanced Fitness Training Group (Active Comparator): This group will receive LEFT with the enhanced Transfer Package (eTP)
  Interventions: Behavioral: Lakeshore Enriched Fitness Training (LEFT); Behavioral: enhanced Transfer Package (eTP)

INTERVENTIONS:
Behavioral: Constraint-Induced Movement Therapy (CIMT) — Constraint-Induced Movement Therapy (CIMT) is a form of physical rehabilitation based on basic research in behavioral psychology and behavioral neuroscience. The therapy will be given on an outpatient basis for 3.5 hours/day for 10 consecutive weekdays. This treatment has four components: 1. intensive training in use of the more-affected arm; 2. organization of this training following shaping principles, which involve frequent positive feedback and progressively increasing the demand of the task in small increments; 3. discouraging use of the less-affected arm by placing the hand in a padded safety mitt, and 4. a set of behavioral procedures, known as the Transfer Package, for transferring gains from the treatment to real-world setting. In this study, two forms of the Transfer Package, standard and enhanced, will be used and form a separate factor (see below).
  Other Names: CI therapy
  Arms: Enhanced CI Therapy Group; Standard CI Therapy Group
Behavioral: Lakeshore Enriched Fitness Training (LEFT) — This treatment will given on an outpatient basis for 3.5 hours per day for 10 consecutive weekdays. It will consist of the following components: general fitness exercises (largely lower extremity), sports and recreation (land and water-based); adapted Yoga; breathing exercises and postural control, movement to music, massage therapy, meditation and Progressive Muscle Relaxation (PMR).
  Arms: Enhanced Fitness Training Group; Standard Fitness Training Group
Behavioral: standard Transfer Package (sTP) — This intervention will take, on average, 30 minutes out of the 3.5 hour daily planned for treatment. The sTP is a set of behavioral procedures for transferring gains from the treatment setting to real-world. The procedures when the sTP is applied to CIMT include negotiating a behavioral contract with the patient and caregiver, when available, about use of each arm during the treatment period, keeping a daily diary on arm use, completing a structured interview about use of the more-affected arm in daily, problem solving about perceived barriers to use of the more-affected arm outside the treatment setting during treatment, and four weekly follow-up phone calls to assess use of the more-affected arm and problem solve about any remaining barriers perceived to its use. The sTP when applied to the LEFT intervention will have parallel components that target engagement in fitness activities and overcoming perceived barriers to fitness in the home.
  Arms: Standard CI Therapy Group; Standard Fitness Training Group
Behavioral: enhanced Transfer Package (eTP) — This intervention will take, on average, 30 minutes out of the 3.5 hour daily planned for treatment. It is an enhanced form of the sTP. The enhancements include a computerized version of the daily diary, cues to be placed in patients' homes to prompt engagement in desired activities, and additional follow-up phone calls.
  Arms: Enhanced CI Therapy Group; Enhanced Fitness Training Group

SUMMARY:
The purpose of this study is to determine the value of Constraint-Induced Movement therapy (CIMT) for improving motor function and general fitness in adults with subacute and chronic traumatic brain injury (TBI), particularly TBI acquired during active military duty, in comparison to a Lakeshore Enriched Fitness Training (LEFT). The study will also test the effect of a set of enhanced versus "standard" procedures for transferring therapeutic gains from treatment setting to everyday life. Lastly, this study will determine whether any therapeutic effects observed are correlated with neuroplastic white matter or grey matter changes.

DETAILED DESCRIPTION:
The proposed project is a prospective, randomized, controlled, single-blind study comparing the motor improvements resulting from Constraint-Induced Movement Therapy (CIMT) and Lakeshore Enriched Fitness Training (LEFT) for traumatic brain injury (TBI) in veterans and civilians. Over the course of two years, there will be a total of 80 subjects randomly assigned to 4 conditions. Treatment, testing, and follow-up testing will be carried out in the first 3 grant years and the 1-year follow-up will be completed in the fourth year. Clinical testing will be conducted at pre-treatment, post-treatment, and 1-year follow-up. Longitudinal neuroimaging studies to determine the treatment change in white matter, grey matter, and functional brain connectivity will be carried out across the above-noted time points by different diffusion tensor imaging (DTI) analysis variants, voxel-based morphometry (VBM) analysis of structural magnetic resonance imaging (MRI) scans, analysis of resting state functional MRI (fMRI), and analysis of fMRI during hand movement.

The 80 study participants will be randomly assigned in equal numbers to 1 of 4 arms: CIMT with Standard Transfer Package (sTP), CIMT with Enhanced Transfer Package (eTP), LEFT with sTP or LEFT with eTP. Forty volunteers will be tested on average per year. The patients will be classified into mild/moderate (Grade 2) and moderate motor deficits (Grades 3); a classification made at the impairment level based on standard active range of motion (AROM) criteria (further elaborated in "Eligibility Criteria").

The primary clinical outcome will be pre- to post-treatment change in a measure of use of the more-affected arm in daily life known as the Motor Activity Log. It is described in the outcomes section. As noted above, the response of the brain to the interventions will be examined using structural grey matter MRI analysis, DTI, and fMRI during resting state and during arm movement.

Each participant will have the option of being accompanied by a caregiver (travel and living expenses paid for by the project). The caregiver will be asked to complete the MAL independently of the participant. The same questionnaire administered to the patient will be administered to the caregiver. In addition, the caregiver will be shown how to help the patient carry out the home practice exercises so that they can do this during treatment and afterwards (if they remain in close contact with the participant).

ELIGIBILITY:
Inclusion Criteria:

- Motor criteria will be made using an impairment-level system for characterizing the severity of an upper-extremity (UE) motor deficit based on Active Range of Motion (AROM). All UE motor criteria determinations will be made with the subject sitting. The more-affected forearm will be resting on a supporting surface (e.g. arm of chair) to allow for maximum wrist flexion with gravity. This study will treat patients at levels of Grade 2 (mild/moderate impairment) and Grade 3 (moderate impairment).

* The minimum motor criterion (MMC) for inclusion in Grade 3 (moderate impairment) will be ability to:

  * Extend against gravity at least 10 degrees at the wrist from a fully flexed starting position
  * Extend two or more fingers at least 10 degrees at the metacarpophalangeal (MP) joint and either the proximal or distal interphalangeal (IP) joints
  * Extend or abduct the thumb at least 10 degrees
  * Extend the elbow at least 20 degrees from a 90 degree flexed starting position
  * Flex and abduct the shoulder at least 45 degrees
* The MMC for inclusion in Grade 2 (mild/moderate impairment) will be ability to:

  * Extend against gravity at least 20 degrees at the wrist from a fully flexed starting position
  * Extend all fingers at least 10 degrees at the MP joint and either the proximal or distal IP joints
  * Extend or abduct the thumb at least 10 degrees
  * Extend the elbow at least 20 degrees from a 90 degree flexed starting position
  * Flex and abduct the shoulder at least 45 degrees
* Additionally, subjects must have substantially reduced use of the extremity in the activities of daily living as indicated by a score of less than 2.5 on the Motor Activity Log (MAL).

Note: Each movement described above must be repeated 3 times in 1 minute.

Exclusion Criteria:

* Those < 3 months post-TBI.
* Excessive UE spasticity.
* Insufficient stamina to carry out the requirements of the therapy (based on clinical judgment).
* Medication (including psychoactive substances) will not be exclusionary except in the following cases: (If subjects are on other medications, the medications will be recorded and the possible effect on treatment outcome will be analyzed separately)

  * Participation in any experimental drug field study
  * Botox injections to the more-affected UE less than 3 months prior to participation
  * Baclofen or Dantrium taken orally at the time of study
* Mini-Mental Status Exam (MMSE) score below 20.
* Concurrent participation in any formal physical rehabilitation program or clinical trial.
* Excessive pain in any joint of the more-affected extremity that could limit ability to cooperate with the intervention (based on clinical judgment).
* Serious, uncontrolled medical problems (e.g., cardiovascular, severe rheumatoid arthritis, serious joint deformity of arthritic origin, symptomatic cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, uncontrolled epilepsy) as judged by the Medical Director.
* Other neurological or musculoskeletal conditions affecting UE function.
* Unable to read or speak English.
* Inadequate communication skills, i.e., not able to reliably understand questions or not able to express needs or report own behavior, to participate in study based on clinical judgment.
* Substantial use of the more-affected arm in daily life as reflected by a Motor Activity Log score > 2.5.
* Pain that interferes with use of the more-affected arm based on clinical judgment.
* A positive pregnancy test will exclude participants from MRI scanning, but would not exclude them from clinical treatment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-09; Primary Completion 2018-01 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Motor Activity Log | From baseline to 19 days
  The Motor Activity Log (MAL) is a structured interview intended to examine how much and how well the subject uses their more-affected arm outside of the laboratory setting.

SECONDARY OUTCOMES:
Accelerometry | From baseline to 19 days
  Accelerometers are devices that monitor movement. Here, they will be worn on the wrist and measure amount of arm movement and overall physical activity.
Accelerometry | From baseline to 12-months
  Accelerometers are devices that monitor movement. Here, they will be worn on the wrist and measure amount of arm movement and overall physical activity.
Motor Activity Log | From baseline to 12-months
  See description of MAL under primary outcome measure.
Six-Minute Walk/Push Wheelchair Test | From baseline to 19 days
  This is a standard test of endurance and physical fitness. The distance walked or wheelchair is pushed in 6 minutes is measured.
Six-Minute Walk/Push Wheelchair Test | From baseline to 12-months
  This is a standard test of endurance and physical fitness. The distance walked or wheelchair is pushed in 6 minutes is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Taub, Ph.D., Principal Investigator — CI Therapy Research Group and Taub Training Clinic
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via FITBIR site after trial has been unblinded and key outcome papers have been published.

REFERENCES:
- [Background] Taub E, Miller NE, Novack TA, Cook EW 3rd, Fleming WC, Nepomuceno CS, Connell JS, Crago JE. Technique to improve chronic motor deficit after stroke. Arch Phys Med Rehabil. 1993 Apr;74(4):347-54. PMID 8466415
- [Background] Taub E, Uswatte G, King DK, Morris D, Crago JE, Chatterjee A. A placebo-controlled trial of constraint-induced movement therapy for upper extremity after stroke. Stroke. 2006 Apr;37(4):1045-9. doi: 10.1161/01.STR.0000206463.66461.97. Epub 2006 Mar 2. PMID 16514097
- [Background] Shaw SE, Morris DM, Uswatte G, McKay S, Meythaler JM, Taub E. Constraint-induced movement therapy for recovery of upper-limb function following traumatic brain injury. J Rehabil Res Dev. 2005 Nov-Dec;42(6):769-78. doi: 10.1682/jrrd.2005.06.0094. PMID 16680614
- [Derived] Morris DM, Taub E, Mark VW, Liu W, Brenner L, Pickett T, Stearns-Yoder K, Bishop-McKay S, Taylor A, Reder L, Adams T, Rimmer J, Dew D, Szaflarski J, Womble B, Stevens L, Rothman D, Uswatte G. Protocol for a Randomized Controlled Trial of CI Therapy for Rehabilitation of Upper Extremity Motor Deficit: The Bringing Rehabilitation to American Veterans Everywhere Project. J Head Trauma Rehabil. 2019 Jul/Aug;34(4):268-279. doi: 10.1097/HTR.0000000000000460. PMID 30608308